CLINICAL TRIAL: NCT02400268
Title: Phase 4, Randomized, Controlled Multicentric, Open-label Clinical Trial to Prove That the 7 Day Course of Treatment for Enterobacteriaceae Bacteremia is More Efficient and Equally Safe Than 14 Day Scheme
Brief Title: Antibiotic Treatment Duration (7 vs 14 Days) Comparison in Blood Stream Infection Causes by Enterobacteriaceae
Acronym: SHORTEN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHORTEN
Record Dates: First submitted 2014-08-05; First posted 2015-03-27 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Enterobacteriaceae Infections; Bloodstream Infection
Keywords: Enterobacteriaceae; Bloodstream; Bacteremia; Recurrence; Reinfection
MeSH Terms: conditions — Enterobacteriaceae Infections; Sepsis; Bacteremia; Recurrence; Reinfection | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 7 days course of antibiotic treatment (Experimental): Accepted antibiotic indicated for enterobacteriaceae infections, according to sensibility test performed and daily practice protocols or local guidelines.
  Interventions: Other: 7 days course of antibiotic treatment
- 14 days course of antibiotic treatment (Active Comparator): Accepted antibiotic indicated for enterobacteriaceae infections, according to sensibility test performed and daily practice protocols or local guidelines.
  Interventions: Other: 14 days course of antibiotic treatment

INTERVENTIONS:
Other: 7 days course of antibiotic treatment — Standard antibiotic treatment approved for enterobacteraciae infections
  Other Names: Antibiotics with approved indication
  Arms: 7 days course of antibiotic treatment
Other: 14 days course of antibiotic treatment — Standard antibiotic treatment approved for enterobacteraciae infections
  Other Names: Antibiotics with approved indication
  Arms: 14 days course of antibiotic treatment

SUMMARY:
The antimicrobial crisis is a real problem. Infections produced by multiresistant bacteria are becoming more and more frequent, and available antimicrobial agents are usually scarce. Reducing the duration of antimicrobial treatments is one of the most efficient measures to control the antibiotic pressure and to optimise the use of these agents.

Bloodstream infections produced by Enterobacteria (EB) are very frequent, but the optimal duration of antibiotics to treat them is unknown, as long as no clinical trials have been specifically developed to answer this question.

Basing on expert opinions, the Infectious Diseases Society pf America (IDSA) recommends the bacteremia by EB secondary to vascular catheter infections to be treated for 7 to 14 days. This represents a variability of up to 100%. No recommendations have been published regarding the duration of treatment of bacteremia from other sources.

The objective of this project is to prove that the 7-day course of treatment for EB bacteremia is more efficient and equally safe than the 14-day scheme.

DETAILED DESCRIPTION:
To achieve theses objectives, we propose this randomized, multicentric clinical trial with a superiority design on the duration of antimicrobial treatment for EB bacteremia in adult patients.

ELIGIBILITY:
Inclusion criteria:

* Adults patients (equal or over 18 years old)
* Primary or secondary bloodstream infection produced by enterobacteriaceae
* Source of bacteremia properly controlled or expect to be properly controlled in the next 24 hours (i.e. bacteremia produced by infected vascular catheter, abscess, obstruction of the biliary or urinary tract).
* Patients able to understand the objectives of the clinical trial and informed consent signed.

Exclusion Criteria:

* Pregnancy
* Post-chemotherapy neutropenia expected to persist more than 7 days.
* Source of bacteremia uncontrolled at inclusion period or in the following 24 hours. The source will be considered as uncontrolled if the bacteremia is secondary to a suppurative infection potentially removable, if no action has been taken to eradicate it, including: bacteremia by vascular not removed catheter, cholangitis secondary to not derived obstruction of the biliary tract, deep abscess not drained, pyohydronephrosis without derivation of the urinary tract.
* Bacteremia secondary to infective endocarditis, bone and joint infections, or neurosurgical infections, which may require prolonged antimicrobial therapy
* Bacteremia due to enterobacteriaceae resistant to carbapenemics.
* Polymicrobial bacteremia including microorganisms different to enterobacteriaceae.
* Patients with no expectations of survival in the next 48 hours of inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2014-09; Primary Completion 2016-12-02 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Days of antimicrobial treatment | 28 days
  To prove that 7-days course of antibiotic therapy is more efficient than 14-days course when treating Enterobacteriaceae bacteremia, in terms of number of days at the end of follow up.

SECONDARY OUTCOMES:
Adverse reactions related to antimicrobial treatment | 28 days
  To prove that 7-days course of antibiotic therapy is as safe as a 14-days course in terms of : Rate of adverse effects including: adverse reactions to drugs, superinfections by resistant bacteria or diarrhea by Clostridium difficile, mortality, relapse of the infection
Cure of bacteremia | 28 days
  Clinical and microbiological cure
Procalcitonin levels | 7-days and 14-days
  To analyze the utility of procalcitonin as a biomarker to decide the end of the antimicrobial treatment of Enterobacteriaceae bacteremia

CONTACTS AND LOCATIONS:
Overall Officials: Jose Molina Gil-Bermejo, MD. PhD, Study Director — Hospitales Universitarios Virgen del Rocío
Locations (4):
- Spain (4):
  - University Hospital Reina Sofía, Córdoba, Córdoba
  - Universitary Hospital Málaga, Málaga, Málaga
  - University Hospital Virgen Macarena, Seville, Seville
  - Hospital Universitario Virgen del Rocío, Seville, Seville

IPD SHARING:
Plan to Share IPD: Yes
Anonimized data for primary and secondary variables is planned to be shared with all the participants within 6 months of data completion.

REFERENCES:
- See also: This organization is formed by 16 Spanish leading research groups in the field, is public funded by Spanish Carlos III Institute and co-financed by European Development Regional Fund (ERDF) — http://www.reipi.org/